CLINICAL TRIAL: NCT04172740
Title: Assessment of Skin Quality Parameters Following RADIESSE Injection in Perioral and Marionette Lines
Brief Title: RADIESSE Injection in Perioral and Marionette Lines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-VP-003R
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Skin Quality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Radiesse (calcium hydroxylpatite)

INTERVENTIONS:
Device: Radiesse (calcium hydroxylpatite) — RADIESSE® injectable implant is a sterile, non-pyrogenic, semi-solid, cohesive implant, whose principle component is synthetic calcium hydroxylapatite (CaHA) suspended in a gel carrier of sterile water for injection, glycerin and sodium carboxymethylcellulose. RADIESSE injectable implant has a CaHA particle size range of 25-45 microns. RADIESSE is available in 1.5cc and 0.8cc pre-filled syringes.
  RADIESSE injectable implant is indicated for subdermal implantation for the correction of moderate to severe facial wrinkles and folds, such as nasolabial folds and it is also intended for restoration and/or correction of the signs of facial fat loss (lipoatrophy).

SUMMARY:
Following treatment with Radiesse, many patients mention an improvement in skin texture This observation is independent from the improvement observed on their facial shape. There is therefore a need to identify and quantify changes in skin parameters following treatment with Radiesse

ELIGIBILITY:
Inclusion Criteria:

1. At the time of consent, women between the ages of 18 and 80 years old;
2. Patient requires lower face treatment (perioral/marionette region) with RADIESSE;
3. Willingness to comply with study requirements;
4. Provide written consent;
5. Patient has a rating of 2 or 3 at Baseline on the Merz Marionette Grading Scale, as per the investigator;
6. Accepted the obligation not to receive any other facial procedures through the follow-up;
7. Understood and accepted the obligation and would be logistically able to appear for all scheduled follow-up visits;
8. No previous facial fillers for a period of 12 months prior to this study;
9. No previous facial fillers in the lower face for 18 months prior to this study.

Exclusion Criteria:

1. Current Pregnancy or lactation [sexually active women of childbearing age must agree to use medically acceptable methods of contraception for the duration of this study (e.g., oral contraceptives, condoms, intrauterine device, shot/injection, patch)];
2. Hypersensitivity to RADIESSE, calcium hydroxylpatite filler or local anesthetics;
3. Patient has received any lower face treatment during the last 12 months, or neuromodulator in the last 6 months;
4. Patient has received mentalis muscle injections of any kind (BoNT-A or fillers) in the last 6 months;
5. Patients meeting any official RADIESSE contra-indications;
6. Patients presenting with porphyria;
7. Inability to comply with follow-up and abstain from facial injections during the study period;
8. Heavy smokers, classified as smoking more than 12 cigarettes per day;
9. History of severe or multiple allergies manifested by anaphylaxis;
10. Previous tissue revitalization therapy in the treatment area within 6 months before treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling, or dermabrasion;
11. Previous surgery including aesthetic facial surgical therapy or liposuction, piercing, or tattoos in the treatment area;
12. History or presence of any disease or lesion near or at the treatment area, including inflammation, active or chronic infection, including in the mouth, dentals, head and neck region;
13. Facial psoriasis, eczema, acne, rosacea, perioral dermatitis and herpes zoster in the treatment area;
14. Cancer or precancer in the treatment area, e.g. actinic keratosis;
15. History of bleeding disorders or treatment with thrombolytics, anticoagulants, or inhibitors of platelet aggregation (e.g. Aspirin or other non-steroid anti-inflammatory drugs [NSAIDs]), within 2 weeks before treatment;
16. Patients using immunosuppressants;
17. Patients with a tendency to form hypertrophic scars or any other healing disorders;
18. Patients with known hypersensitivity to lidocaine or agents structurally related to amide type local anaesthetics (e.g., certain anti-arrhythmics);
19. Patients administered dental block or topical administration of lidocaine;
20. Patients with epilepsy, impaired cardiac conduction, severely impaired hepatic function or severe renal dysfunction.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-11 (Actual)

PRIMARY OUTCOMES:
Hydration | Month 3
  Assessment of changes in hydration at Month 3, as assessed with the Courage and Khazaka system device, following the injection of RADIESSE, in perioral and marionette lines regions

SECONDARY OUTCOMES:
Hydration | Month 6
  Changes in hydration at Month 6, as assessed with the Courage and Khazaka system device;
Elasticity | Month 3 and 6
  Changes in elasticity at Month 3 and 6, as assessed with the Courage and Khazaka system device;
pH | Month 3 and 6
  Changes in pH and quality of skin barrier function (TEWL - Trans Epidermal Water Loss) at Months 3 and 6, as assessed with the Courage and Khazaka sys
Skin texture | Month 3 and 6
  Changes in skin surface textural irregularities, smoothness, roughness, wrinkles and scaliness) at Months 3 and 6, as assessed with the Courage and Khazaka system.
Merz validated marionette scale | Month 3 and 6
  Changes in the aesthetic improvement using the Merz validated marionette scale at Months 3 and 6. This is a 5-point scale, where 0 = no lines and 4 = very severe lines.
Global Assessment Improvement Scale | Months 3 and 6
  Changes in the aesthetic appearance using the Global Assessment Improvement Scale (GAIS) using standardised 2D/3D photographs for patients and blinded physicians at Months 3 and 6;
Fitzpatrick Wrinkle Assessment Scale | Months 3 and 6
  1. Changes in skin quality using the modified Fitzpatrick Wrinkle Assessment Scale (FWAS) and standardised 2D/3D photographs at Months 3 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, FRCSC, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc, Montreal, Quebec, Canada